CLINICAL TRIAL: NCT06781996
Title: Phase III Randomized Controlled Open Label Clinical Trial to Determine the Efficacy of a Digital Self-management Support Tool to Improve the Quality of Life During Adjuvant HOrmonal Therapy for Patients With Early Breast Cancer
Brief Title: A Study to Determine the Efficacy of a Digital Self-management Support Tool to Improve the Quality of Life During Adjuvant HOrmonal Therapy for Patients With Early Breast Cancer
Acronym: HOPE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Resilience (Industry); WeShare (Unknown); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-A01127-40; 2024/3897 (Other: CSET number)
Record Dates: First submitted 2024-12-31; First posted 2025-01-17 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: early stage breast cancer; Hormone-receptor positive; endocrine therapy-related adverse events
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized trial that compares a personalized digitally-enabled pathway delivered by a mobile application in addition to standard of care vs. standard of care alone in patients with HR+ early breast cancer reporting endocrine therapy-related adverse events.
  The HOPE study is a national, prospective, randomized, open-label trial conducted in France. 180 patients will be randomly assigned 1:1 to receive either 12 weeks of multimodal Resilience© digital companion including education and self-care modules in addition to the standard of care provided by their treating oncologists and supportive care team at their care centers or 12 weeks of standard of care provided by their treating oncologists and supportive care team at their care centers.
  Data from the literature in oncology trials with Patient-Reported Outcomes suggests that in the absence of double-blind concealment, clinically important differences could still be detected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard supportive care and multimodal Resilience© digital companion with digital self care program (Experimental): Patients will receive standard of care provided by the oncologist and supportive care team at the patient local cancer center including referrals for local supportive care programs. In addition, patients will have access to Resilience© a multi-component, multi-level interventional mobile application that will offer: (a) supportive educational care information (b) self-symptom management resources with availability of a remote health-care provider evaluation that addresses patient-specific needs in survivorship care and recommends personalized digital self-management resources at onboarding and if needed in case of low engagement in the mobile app.
  Interventions: Other: multimodal Resilience© digital companion; Other: Standard supportive care
- Standard supportive care (Active Comparator): Patients will receive standard of care provided by the oncologist and supportive care team at the patient local cancer center including referrals for local supportive care programs. Local supportive care programs may also include the use of already deployed remote patient monitoring and solutions, digital and in person education.
  Interventions: Other: Standard supportive care

INTERVENTIONS:
Other: multimodal Resilience© digital companion — Resilience© is a multi-component, multi-level interventional mobile application that will offer: (a) supportive educational care information (b) self-symptom management resources with availability of a remote health-care provider evaluation that addresses patient-specific needs in survivorship care and recommends personalized digital self-management resources at onboarding and if needed in case of low engagement in the mobile app.
  Intervention duration : 3 weeks
  Arms: Standard supportive care and multimodal Resilience© digital companion with digital self care program
Other: Standard supportive care — standard of care provided by the oncologist and supportive care team at the patient local cancer center including referrals for local supportive care programs. Local supportive care programs may also include the use of already deployed remote patient monitoring and solutions, digital and in person education.

SUMMARY:
Randomized trial that compares a personalized digitally-enabled pathway delivered by a mobile application in addition to standard of care vs. standard of care alone in patients with HR+ early breast cancer reporting endocrine therapy related adverse events.

The HOPE study is a national, prospective, randomized, open-label trial conducted in France. 180 patients will be randomly assigned 1:1 to receive either 12 weeks of multimodal Resilience© digital companion including education and self-care modules in addition to the standard of care provided by their treating oncologists and supportive care team at their care centers or 12 weeks of standard of care provided by their treating oncologists and supportive care team at their care centers.

Data from the literature in oncology trials with Patient-Reported Outcomes suggests that in the absence of double-blind concealment, clinically important differences could still be detected.

ELIGIBILITY:
Inclusion Criteria:

1. Documentation of Disease:

   1. Subjects must have histologically confirmed ER and/or PgR positive HR+ invasive BC;
   2. Subjects must have stage I to III breast cancer and no evidence of distant metastatic or locally recurrent disease;

   NB: Bilateral breast carcinoma is allowed;

   NB: Patients with personal history of previous breast cancer or Ductal Carcinoma in situ (DCIS) are eligible for the protocol;
2. Indication to receive adjuvant endocrine therapy (tamoxifen or aromatase inhibitors) with or without targeted agents (e.g., CDK 4/6 inhibitors, PARP inhibitors, bisphosphonates);
3. Prior treatment: Patients must be actively on ET for their breast cancer diagnosis (any type, including either tamoxifen or an aromatase-inhibitor with or without targeted agents) at the time of study enrollment;
4. Documentation of side effects of ongoing ET: Any endocrine therapy related adverse effects should be reported during treatment with endocrine therapy;
5. Others:

   1. Age ≥ 18 years;
   2. ECOG Performance Status 0,1 or 2;
   3. Patients should possess a smartphone;
   4. Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed;
   5. Patient should be able and willing to comply with study visits and procedures as per protocol;
   6. Patients must be affiliated to a social security system or beneficiary of the same;
   7. Able to readily read and understand French;

NB: Patients may have breast reconstruction during protocol participation;

NB: Biologic therapy, targeted therapy and bisphosphonates are acceptable during protocol participation;

NB: Male patients can be included in the trial;

NB: Pharmacological or other non-pharmacological interventions for endocrine treatment for adverse effects are accepted at physician discretion.

Exclusion Criteria:

1. Severe cognitive impairments or severe psychiatric disorders (assessed by the investigator or mentioned in the medical file of the patient) which in the investigator's opinion would jeopardize compliance with the protocol;
2. Patient under guardianship or deprived of her/his liberty by a judicial or administrative decision or incapable of giving her/his consent;
3. Patients participating at enrollment in a behavioral interventional trial;
4. Patients suffering from physical related reversible and treatable causes of the entry endocrine therapy-related adverse events (e.g. but not limited to anemia, electrolytes unbalance, infections, renal dysfunction, active metastases hormonal unbalances [hypothyroidism, adrenal insufficiency, etc.] - according to physician's judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy of a personalized approach, consisting of a multi-component, interventional mobile application in addition to standard of care, compared with standard care alone in improving quality of life (QOL) after 12 weeks. | up to 12 weeks of intervention
  The primary endpoint of the study is the ET symptoms scale of the European Organization for Research and Treatment of Cancer (EORTC) QOL questionnaire (QLQ)-BR45 over a 12-weeks period.

SECONDARY OUTCOMES:
To evaluate the impact of the intervention on other EORTC QLQ-C30 domains, including fatigue, emotional distress, pain, and sleep quality; | after 12 months of randomization
To evaluate the impact of the intervention on insomnia measured by a wearable device; | up to 12 months after randomization
  Insomnia by a wearable device capturing sleep quality and sleep cycle (Withings© Pulse HR smartwatch);
To evaluate the impact of the intervention on adherence to endocrine therapy, assessed through the modified MIS-A questionnaire | up to 12 months after randomization
  reliable, easy-to-use, self-administered questionnaire, validated in France that is able to longitudinally capture granular data on non-adherence to chronic medication over short and long time.
To evaluate the impact of the intervention on the perceived self-efficacy of symptom management; | up to 12 months after randomization
  Perceived self-efficacy in symptom management will be evaluated using the PROMIS Self-Efficacy for Managing Chronic Conditions - Managing Symptoms - Short Form 8a questionnaire.
To evaluate the impact of the intervention on eHealth Literacy levels | up to 12 months after randomization
  Ability of the patients to find, understand and use information to improve their health from electronic sources using the eHLQ questionnaire
To evaluate the implementation process including the adoption of the HOPE digitally enabled supportive care pathway (Resilience mobile application) | up to 12 weeks of intervention
  Information on digital health adoption and implementation process will be measured by different criteria:
  - Willingness rate (Resilience© digital companion): will be defined as the rate of patients that activated a Resilience account adoption rate (Resilience© digital companion): will be defined as the rate of users who used Resilience as intended Full digital usage experience: using the experience questionnaire developped for the study
To evaluate the patient experience in using a web platform (WeShare) for collecting ePROs data. | up to 12 weeks of intervention
  Using the experience questionnaire developped for the study and the French System Usability Scale
To evaluate the impact of the intervention on physical activity levels measured by a wearable device; | up to 12 weeks of intervention
  Physical activity levels will be captured through a wearable device (number of steps, distance in Km and calories burned) (Withings © Pulse HR smartwatch)

CONTACTS AND LOCATIONS:
Overall Officials: Ines VAZ-LUIS, MD, Study Director — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, France